CLINICAL TRIAL: NCT02605304
Title: Phase II Trial of Retreatment Strategies for Difficult-to-Treat Hepatitis C Virus (HCV)-Infected Individuals Who Have Failed Prior Direct Acting Antiviral (DAA)-Based Regimens
Brief Title: 12 Weeks of Ledipasvir (LDV)/Sofosbuvir (SOF) With Weight-based Ribavirin vs. 24 Weeks of LDV/SOF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study experienced enrollment difficulties.
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5348; UM1AI068636 (NIH)
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: HIV-1 Infection; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: LDV/SOF + RBV (Experimental): Ledipasvir/sofosbuvir + ribavirin for 12 weeks, followed by 24 weeks of post-treatment follow-up.
  Interventions: Drug: Ledipasvir/sofosbuvir; Drug: Ribavirin
- Arm B: LDV/SOF (Experimental): Ledipasvir/sofosbuvir for 24 weeks, followed by 24 weeks of post-treatment follow-up.
  Interventions: Drug: Ledipasvir/sofosbuvir

INTERVENTIONS:
Drug: Ledipasvir/sofosbuvir — Participants were prescribed one fixed dose tablet of LDV 90 mg/SOF 400 mg orally per day.
  Other Names: LDV/SOF; Harvoni
Drug: Ribavirin — Based on weight at entry:
  For weight <75 kg, participants were prescribed 1000 mg of RBV per day, divided into two doses to be taken orally.
  For weight ≥75 kg: participants were prescribed 1200 mg of RBV per day, divided into two doses to be taken orally.
  Other Names: RBV
  Arms: Arm A: LDV/SOF + RBV

SUMMARY:
People who are infected with Hepatitis C Virus (HCV) have a great chance of being cured of the infection when they are treated with sofosbuvir. However, in some instances, treatment with sofosbuvir-containing therapy does not work. It is not known if people respond to retreatment with sofosbuvir, after it did not work the first time. There is an important need to understand retreatment options in those instances. This clinical trial was done to study the response to two different regimens, ledipasvir/sofosbuvir and ledipasvir/sofosbuvir with ribavirin, and to see if they are safe and well-tolerated in HCV-infected persons whose previous treatment with sofosbuvir had failed.

DETAILED DESCRIPTION:
There is a pressing need to understand appropriate retreatment options for HCV-infected patients who fail direct acting antiviral (DAA)-based regimens. To date, over 100,000 prescriptions have been written for SOF. Recent data indicate that SOF-based treatment defined as SOF/RBV, SOF/pegylated-interferon (PEG-IFN)/RBV or SOF/simeprevir (SIM) +/- RBV have led to treatment response of 70-92% in HCV genotype (GT) 1 patients, depending on the regimen used and presence of liver cirrhosis. Thus, there is a growing number of individuals who have failed SOF-based regimens and are in need of a retreatment strategy, the majority of which are anticipated to be HCV GT1, given the US distribution of genotypes. There are no data to inform retreatment strategies for HIV-infected individuals with SOF failure, who have traditionally represented a harder to treat group and are impacted by DAA-antiretroviral (ARV) interactions.

This was a phase II retreatment study of HCV GT1 and HIV coinfected participants who had previous HCV virologic failure on a SOF-based regimen. Participants were randomized to one of two treatment arms: 12 weeks of LDV/SOF with weight-based RBV (Arm A) or 24 weeks of LDV/SOF alone (Arm B). The targeted sample size was 40, 20 participants in each arm.

Post-entry, the study visits were scheduled at weeks 1, 2, 4, 8, 12, 16, 20 and 24 after study entry (with week 16, 20, 24 visits limited to those on the 24-week regimen), and at 4, 12 and 24 weeks after treatment discontinuation. The total study duration was 36 weeks in Arm A and 48 weeks in Arm B. At each visit, a physical examination and blood collection were conducted. HCV RNA was tested at each visit. For female participants of reproductive potential, pregnancy tests were done. At on-treatment visits, participants also completed an HCV treatment adherence questionnaire. Urinalysis was conducted at all on-treatment visits and at 4 weeks post treatment. At select visits, plasma, whole blood, urine and dried blood spots were collected.

The study was randomized because there was clinical equipoise on the benefits and drawbacks in the two study arms. The study was not designed to be powered for comparisons between the randomized study arms, and no formal statistical comparisons were conducted. The primary analysis was conducted as a single-arm analysis for each regimen.

The study experienced enrollment difficulties due to the small number of HCV treatment failures from select SOF-based regimens who would be eligible for this study, and closed to accrual prematurely. The participants enrolled remained on study until completion of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Documentation of non-cirrhotic or cirrhotic status
* HIV-1 infection
* HIV antiretroviral treatment status (ART), CD4+ T-cell (CD4) count and HIV-1 RNA as follows: (1) not on ART with CD4 count >500 cells/mm^3 within 42 days of study entry, (2) elite controller not on ART with CD4 >200 cells/mm^3 within 42 days of study entry and HIV-1 RNA <500 copies/mL on all measurements within 48 weeks prior to study entry, (3) on a stable protocol-approved ART with CD4 count >200 cells/mm^3 and HIV-1 RNA <50 copies/mL within 42 days of study entry
* HCV GT-1 within 12 months prior to study entry
* Prior virologic treatment failure with SOF-containing regimen (SOF/RBV, SOF/PEG/RBV, and SOF/SIM)
* Body mass index (BMI) ≥18 kg/m^2 within 42 days prior to study entry
* Certain laboratory values obtained within 42 days prior to study entry
* Hemoglobin ≥12.0 g/dL for male, ≥11.0 g/dL for female participants
* Aspartate aminotransferase (AST) (SGOT) and Alanine aminotransferase (ALT) (SGOT) <10 x ULN
* For female participants of reproductive potential, a negative serum pregnancy test with a sensitivity of at least 25 mIU/mL performed at screening and within 48 hours prior to study entry
* Agreement to use at least two reliable forms of contraceptive simultaneously while receiving study treatment and for 6 months afterward
* Intention to comply with the dosing instructions and study schedule of assessments

Exclusion Criteria:

* Receipt of any investigational drug or device within 60 days prior to study entry
* Prior exposure to a DAA other than SOF and SIM
* Chronic liver disease of a non-HCV etiology
* Presence of active or acute AIDS-defining opportunistic infections within 42 days prior to study entry
* Active, serious infection (other than HIV-1 or HCV) requiring parenteral antibiotics, antivirals, or antifungals within 42 days prior to study entry
* Hepatitis B virus (HBV) infection (defined as HBsAg positive) within 42 days prior to study entry
* History of clinically significant hemoglobinopathy
* Chronic current use of systemically administered immunosuppressive agents
* History of solid organ transplantation
* Current or prior history of clinical hepatic decompensation
* History of a gastrointestinal disorder (or postoperative condition) that could interfere with the absorption of the study drug
* History of significant or symptomatic pulmonary disease, cardiac disease, or porphyria that in the opinion of the investigator would interfere with the study
* History of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
* Active drug or alcohol use or dependence
* Use of any prohibited concomitant medications per the LDV/SOF product labeling, within 42 days prior to study entry
* Known hypersensitivity to RBV, SOF, LDV, their metabolites, or formulation excipients or any other contraindication to the use of RBV, SOF or LDV
* Currently receiving zidovudine (ZDV), didanosine (ddI), stavudine (d4T) or tipranavir
* Acute HIV infection defined as the phase immediately following infection during which anti-HIV antibodies are undetectable
* Known hepatocellular carcinoma
* Breastfeeding or pregnancy
* A male participant with a pregnant female partner
* Receipt of colony stimulating agents, including but not limited to erythropoietin, within 42 days prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Luetkemeyer, MD, Study Chair — University of California, San Francisco HIV/AIDS CRS; Jennifer J. Kiser, PharmD, Study Chair — University of Colorado, Denver
Locations (2):
- United States (2):
  - Ucsf Aids Crs (801), San Francisco, California
  - 7804 Weill Cornell Chelsea CRS, New York, New York

REFERENCES:
- [Result] Tam E, Luetkemeyer AF, Mantry PS, Satapathy SK, Ghali P, Kang M, Haubrich R, Shen X, Ni L, Camus G, Copans A, Rossaro L, Guyer B, Brown RS Jr; RESCUE and ACTG A5348 study investigators. Ledipasvir/sofosbuvir for treatment of hepatitis C virus in sofosbuvir-experienced, NS5A treatment-naive patients: Findings from two randomized trials. Liver Int. 2018 Jun;38(6):1010-1021. doi: 10.1111/liv.13616. Epub 2017 Dec 5. PMID 29091342
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf?sfvrsn=8
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.tech-res.com/docs/default-source/safety/manual_for_expedited_reporting_aes_to_daids_v2.pdf?sfvrsn=12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February to June 2016 at 3 U.S. sites.
Period: Overall Study
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [49 to 57] | 58 [49 to 65] | 53 [49 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 7
Intravenous drug use history [Count of Participants; unit: Participants]
  Never | 2 | 3 | 5
  Previously | 2 | 0 | 2
Prior hepatitis C virus (HCV) treatment regimen [Count of Participants; unit: Participants]
  SOF/RBV | 2 | 1 | 3
  SOF/RBV/PEG-IFN | 2 | 2 | 4
Cirrhosis status [Count of Participants; unit: Participants] — Cirrhotic was defined as: liver biopsy showing cirrhosis (Metavir score =4, Ishak score ≥5 or equivalent) at any time prior to study entry; or transient elastography (FibroScan®; Echosens, Paris, France) ≥12.5 kPa within 12 months of study entry; or HCV FibroSURE® (Laboratory Corporation of America, Raritan, NJ, USA) score of ≥0.72 with aspartate aminotransferase:platelet ratio index (APRI) ≥2 within 12 months of study entry.
  Participants
    Cirrhotic | 1 | 0 | 1
    Non-cirrhotic | 3 | 3 | 6
HCV genotype [Count of Participants; unit: Participants]
  1A | 2 | 3 | 5
  1B | 2 | 0 | 2
HCV RNA [Median (Inter-Quartile Range); unit: log10 IU/mL] — HCV RNA testing was performed at a central laboratory using the COBAS® AmpliPrep/COBAS® TaqMan® HCV Quantitative Test, version 2.0 (Roche Diagnostics, Rotkreuz, Switzerland).
  log10 IU/mL | 6.31 [5.80 to 6.66] | 7.01 [6.73 to 7.48] | 6.71 [6.00 to 7.01]
HIV antiretroviral treatment (ART) status [Count of Participants; unit: Participants]
  On ART | 4 | 3 | 7
  Not on ART | 0 | 0 | 0
HIV-1 RNA quantitation [Count of Participants; unit: Participants] — HIV-1 RNA testing was performed at a central laboratory using Abbott RealTime HIV-1 assay (Abbott Laboratories, Lake Bluff, IL, USA). Unquantifiable was defined as below the lower limit of quantitation (LLOQ) of the assay (40 copies/mL).
  Participants
    Unquantifiable | 4 | 3 | 7
    Quantifiable | 0 | 0 | 0
CD4+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 564 [435 to 614] | 387 [200 to 1150] | 528 [341 to 628]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks After Treatment Discontinuation (SVR12)
Description: SVR12 was defined as HCV RNA below the LLOQ of the assay (either target detected [TD] or target not detected [TND]) at 12 weeks after treatment discontinuation. The sample within the visit window, closest to the targeted time was used. If there was no HCV RNA sample within visit window, then the participant was considered not to have achieved SVR12, unless there were preceding and subsequent HCV RNA measurements that were both <LLOQ (either TD or TND). HCV RNA testing was conducted at a central laboratory using the COBAS® AmpliPrep/COBAS® TaqMan® HCV Quantitative Test, version 2.0 (Roche Diagnostics, Rotkreuz, Switzerland). Wilson (score) method was used for confidence intervals.
Time Frame: At 12 weeks after treatment discontinuation (i.e., at 24 weeks after study entry in Arm A and at 36 weeks after study entry in Arm B).
Population: All participants enrolled.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
percentage of participants | 100.0 [59.7 to 100.0] | 100.0 [52.6 to 100.0]

2. Primary Outcome: Percentage of Participants With Grade 3 or Higher Adverse Event (AE), Serious AE (SAE), or AE Reported as the Reason for Permanent Discontinuation of Study Treatment
Description: Percentage of participants who experienced an AE (diagnosis, sign/symptom or laboratory abnormality) of ≥Grade 3, SAE according to International Conference on Harmonisation (ICH) criteria, or AE reported as the reason for permanent study treatment discontinuation, during study treatment and up to 30 days after study treatment. Events that were ongoing at the same grade from prior to study treatment initiation were excluded. AEs were graded by the clinicians according to the Division of AIDS (DAIDS) AE Grading Table (V2.0) as follows: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-Threatening. The percentage of participants who experienced any event (overall), and the percentage of participants who experienced each component of the outcome are provided in the data table below. The categories are not mutually exclusive. A participant may have experienced multiple events. Each participant is counted at most once within category, and in the overall summary line.
Time Frame: From study treatment initiation to 30 days after study treatment discontinuation. Duration of treatment was 12 weeks in Arm A and 24 weeks in Arm B.
Population: All participants enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
percentage of participants
  Overall (any event) | 50.0 | 0
  Diagnosis ≥ Grade 3 | 0 | 0
  Laboratory event ≥ Grade 3 | 50.0 | 0
  Sign/symptom ≥ Grade 3 | 0 | 0
  SAE | 0 | 0
  AE that led to treatment discontinuation | 0 | 0

3. Secondary Outcome: Percentage of Participants With Protocol-specified Renal Events
Description: The study protocol defined renal events as (1) ≥Grade 2 creatinine clearance (CRCL) after study entry, or (2) new urinalysis proteinuria and/or glucosuria, defined as ≥1+ or an increase ≥1+ from baseline. The percentage of participants who experienced any renal event, and the percentages of participants who experienced each component of the outcome are provided in the data table below. The categories are not mutually exclusive. A participant may have experienced multiple events. Each participant is counted at most once within category, and in the overall summary line.
Time Frame: From study entry to study completion (Week 36 in Arm A, Week 48 in Arm B)
Population: All participants enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
percentage of participants
  Overall (any renal event) | 25.0 | 33.3
  CRCL ≥ Grade 2 | 25.0 | 33.3
  Proteinuria | 25.0 | 0
  Glucosuria | 0 | 0

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 Weeks After Treatment Discontinuation (SVR4)
Description: SVR4 was defined as HCV RNA below the LLOQ of the assay (either TD or TND) at 4 weeks after treatment discontinuation. The sample within the visit window, closest to the targeted time was used. If there was no HCV RNA sample within visit window, then the participant was considered not to have achieved SVR4, unless there were preceding and subsequent HCV RNA measurements that were both <LLOQ (either TD or TND). HCV RNA testing was conducted at a central laboratory using the COBAS® AmpliPrep/COBAS® TaqMan® HCV Quantitative Test, version 2.0 (Roche Diagnostics, Rotkreuz, Switzerland). Wilson (score) method was used for confidence intervals.
Time Frame: At 4 weeks after treatment discontinuation (i.e., at 16 weeks after study entry in Arm A and at 28 weeks after study entry in Arm B).
Population: All participants enrolled.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
percentage of participants | 100.0 [59.7 to 100.0] | 100.0 [52.6 to 100.0]

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 24 Weeks After Treatment Discontinuation (SVR24)
Description: SVR24 was defined as HCV RNA below the LLOQ of the assay (either TD or TND) at 24 weeks after treatment discontinuation. The sample from a visit greater than 20 weeks after treatment discontinuation which was closest to the targeted week (24 weeks post treatment), not followed by any HCV RNA result ≥LLOQ, was used. If there was no HCV RNA sample within this window, then the participant was considered not to have achieved SVR24. HCV RNA testing was conducted at a central laboratory using the COBAS® AmpliPrep/COBAS® TaqMan® HCV Quantitative Test, version 2.0 (Roche Diagnostics, Rotkreuz, Switzerland). Wilson (score) method was used for confidence intervals.
Time Frame: At 24 weeks after treatment discontinuation (i.e., at 36 weeks after study entry in Arm A and at 48 weeks after study entry in Arm B).
Population: All participants enrolled.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
percentage of participants | 100.0 [59.7 to 100.0] | 100.0 [52.6 to 100.0]

6. Secondary Outcome: Number of Participants With Unquantifiable HCV RNA
Description: Unquantifiable HCV was defined as HCV RNA below the LLOQ of the assay (15 IU/mL), either TD or TND. HCV RNA testing was conducted at a central laboratory using the COBAS® AmpliPrep/COBAS® TaqMan® HCV Quantitative Test, version 2.0 (Roche Diagnostics, Rotkreuz, Switzerland).
Time Frame: Entry (Week 0); at 1, 4, 8, 12 (and 16, 20, 24 in Arm B) weeks after study entry
Population: All participants enrolled who had HCV RNA results available at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
Participants
  Week 0: unquantifiable HCV RNA | 0 | 0
  Week 1: unquantifiable HCV RNA | 1 | 0
  Week 4: unquantifiable HCV RNA | 4 | 3
  Week 8: unquantifiable HCV RNA | 4 | 3
  Week 12: unquantifiable HCV RNA: number analyzed (Participants) | 4 | 2
  Week 12: unquantifiable HCV RNA | 4 | 2
  Week 16: unquantifiable HCV RNA: number analyzed (Participants) | 0 | 3
  Week 16: unquantifiable HCV RNA |  | 3
  Week 20: unquantifiable HCV RNA: number analyzed (Participants) | 0 | 3
  Week 20: unquantifiable HCV RNA |  | 3
  Week 24: unquantifiable HCV RNA: number analyzed (Participants) | 0 | 3
  Week 24: unquantifiable HCV RNA |  | 3

7. Secondary Outcome: Number of Participants With HIV-1 RNA >50 Copies/mL
Description: HIV-1 RNA testing was performed at a central laboratory using Abbott RealTime HIV-1 assay (Abbott Laboratories, Lake Bluff, IL, USA).
Time Frame: Entry (Week 0); at 4, 12 (and 24 in Arm B) weeks after study entry, and at 4 weeks after treatment discontinuation
Population: All participants enrolled with HIV-1 RNA results available at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
Participants
  Week 0: HIV-1 RNA >50 copies/mL | 0 | 0
  Week 4: HIV-1 RNA >50 copies/mL | 0 | 0
  Week 12: HIV-1 RNA >50 copies/mL: number analyzed (Participants) | 4 | 2
  Week 12: HIV-1 RNA >50 copies/mL | 0 | 0
  Week 24: HIV-1 RNA >50 copies/mL: number analyzed (Participants) | 0 | 3
  Week 24: HIV-1 RNA >50 copies/mL |  | 0
  Post treatment Week 4: HIV-1 RNA >50 copies/mL: number analyzed (Participants) | 4 | 2
  Post treatment Week 4: HIV-1 RNA >50 copies/mL | 0 | 0

8. Secondary Outcome: CD4+ T-cell (CD4) Count Change From Baseline
Description: Change in CD4 count was calculated as value at the post entry visit minus the value at study entry.
Time Frame: Entry and at 12 (and 24 in Arm B) weeks after study entry
Population: All participants enrolled with CD4 result available at entry and at the post-entry visit.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
Number analyzed (Participants) | 4 | 3
cells/mm^3
  Week 12: CD4 change: number analyzed (Participants) | 3 | 2
  Week 12: CD4 change | -102 [-106 to -28] | 365 [196 to 533]
  Week 24: CD4 change: number analyzed (Participants) | 0 | 3
  Week 24: CD4 change |  | 138 [97 to 302]

ADVERSE EVENTS:
Time Frame: From study treatment dispensation to study completion (Week 36 in Arm A, Week 48 in Arm B).
Description: At entry, all diagnoses, signs/symptoms and laboratory values were collected, regardless of grade. Post-entry, diagnoses, signs/symptoms and laboratory values of ≥Grade 3 and events that led to change in treatment (excluding indications for RBV dose modifications) or that met ICH, expedited AE, or SAE guidelines, regardless of grade, were collected. Creatinine and creatinine clearance were reported regardless of grade. The DAIDS AE Grading Table (V2.0) and Expedited AE Manual (V2.0) were used.
Arm/Group | Arm A: LDV/SOF + RBV | Arm B: LDV/SOF
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: LDV/SOF + RBV (N=4) | Arm B: LDV/SOF (N=3)
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Bilirubin conjugated increased (Investigations) | 1 | 1
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase abnormal (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study accrual was terminated prematurely due to enrollment challenges. There was a small number of participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT02605304/SAP_000.pdf
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/04/NCT02605304/Prot_001.pdf